CLINICAL TRIAL: NCT00699179
Title: EFFicacious glycaEmia Control, Treatment Goal achIevement Very simplE With NovoMix 30: A Single-country, Multicentre, Prospective, Open Label, Non-controlled, Observational, 26-week Study in Serbian Patients Using NovoMix® 30 (Biphasic Insulin Aspart 30) for Treatment of Diabetes Mellitus in Everyday Clinical Practice
Brief Title: Observational Study to Evaluate the Efficacy and Safety of NovoMix® 30 in Type 1 and 2 Diabetes
Acronym: EFFECTIVE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3557
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — There is no intervention in this trial. The trial is prepared to be non-interventional one. Start dose and frequency to prescribed by the physician as a result of a normal clinical evaluation.
  Other Names: NovoMix® 30

SUMMARY:
This study is conducted in Europe. This observational study is aimed to reflect the post-authorisation experience with insulin analogue (biphasic insulin aspart 30) when used under normal clinical practice conditions in Serbia.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 Diabetes Mellitus inadequately controlled on human insulin therapy lasting for at least 6 months
* HbA1c greater than 7%
* Informed Consent

Exclusion Criteria:

* Patients with a hypersensitivity to biphasic insulin aspart 30 or to any of the excipients
* Other limiting conditions specified in the locally approved NovoMix 30 SPC ( Summary of Product Characteristics), PIL ( Patient Information Leaflet).
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next couple of months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 and 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 2308 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | After 6 months

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c below 7,5% for Type 1 Diabetes Mellitus, below 7.0% and below or equal to 6.5% for Type 2 Diabetes Mellitus | after 12 weeks and 26 weeks compared to baseline
Change in FPG (glucose variability) | after 12 weeks and 26 weeks compared to baseline
Change in PPG (postprandial control) | after 12 weeks and 26 weeks compared to baseline
Change in insulin dose and number of injections | at 12 weeks and 26 weeks of treatment
Change in oral antidiabetic drug therapy dosage and eventual discontinuation of oral antidiabetic drug therapy during the study | after 12 weeks and 26 weeks of treatment compared to baseline
Change in body weight and waist circumference | at 12 weeks and 26 weeks of treatment compared to baseline
Change in number of major hypoglycaemic events during 4 weeks proceeding routine visits | at 12 weeks and 26 weeks of treatment compared to baseline
Number of adverse drug reactions (ADR) | after 12 weeks and 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Belgrade, Serbia and Montenegro

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com